CLINICAL TRIAL: NCT05383612
Title: To Evaluate the Efficacy of 3% Diquafosol Sodium in the Treatment of Mild to Moderate MGD in Different Treatment Pattern
Brief Title: To Evaluate the Efficacy of Diquafosol Sodium in the Treatment of MGD in Different Treatment Pattern
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Zhongshan Ophthalmic Center, Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Jin Yuan, Professor, Zhongshan Ophthalmic Center, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2022KYPJ085
Record Dates: First submitted 2022-04-13; First posted 2022-05-20 (Actual); Last update posted 2023-02-21 (Actual); Status verified 2023-02

CONDITIONS: Dry Eye; Meibomian Gland Dysfunction
MeSH Terms: conditions — Dry Eye Syndromes; Meibomian Gland Dysfunction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group I:3% diquafosol (Experimental): 70 people, 70 eyes.
  Interventions: Drug: 3% Diquafosol Sodium Eye Drops
- Group II:3% diquafosol and warm compresses and lid massage (Other): 70 people, 70 eyes.
  Interventions: Procedure: Warm compresses; Drug: 3% Diquafosol Sodium Eye Drops

INTERVENTIONS:
Procedure: Warm compresses — Commercial eye patch, 10 min before lid massage.Warm compresses and lid massage every 2 weeks，5 times in total（0，2, 4, 6, 8W）.
  Arms: Group II:3% diquafosol and warm compresses and lid massage
Drug: 3% Diquafosol Sodium Eye Drops — 3% Diquafosol Sodium Eye Drops (DIQUAS ophthalmic solution 3%; Santen Pharmaceutical Co. Ltd, Osaka, Japan)，3% diquafosol was administered six times a day for 12 weeks.

SUMMARY:
MGD is a chronic, diffuse abnormality of the meibomian glands, commonly characterized by terminal duct obstruction and/or qualitative/quantitative changes in the glandular secretion. It may result in alteration of the tear film, symptoms of eye irritation, clinically apparent inflammation, and ocular surface disease. The meibomian glands, found in the upper and lower eyelids, excrete lipids onto the ocular surface that forms the outermost layer of the tear film, lubricating the ocular surface during blinking and protecting against tear evaporation.1 2 Through dysfunction of the meibomian glands, reduced lipid secretion may contribute to tear film instability and entry into the vicious circle of dry eye disease. The prevalence of MGD is higher in Asian populations, ranging from 46% to 70%.

The management and treatment subcommittee of the International Workshop on MGD proposed a treatment algorithm in which treatment is added depending on the severity of MGD. The sequence of treatment addition is eyelid hygiene, eyelid warming and massage, artificial lubricants, topical azithromycin, topical emollient lubricant, oral tetracycline derivatives, lubricant ointment, and anti-inflammatory therapy.

Topical diquafosol solution has been used to treat dry eye because it increases fluid secretion from conjunctival epithelial cells and mucin secretion from conjunctival goblet cells via the P2Y2 receptor. Because P2Y2 receptor expression is observed in sebaceous cells and ductal cells in the meibomian gland, diquafosol is expected to have some effects on meibomian glands. it has been reported that use 3% diquafosol ophthalmic solution in patients with obstructive MGD for more than 4 months. Ocular symptoms, lid margin abnormalities, the superficial punctate keratopathy score, and the meibum grade were decreased, while the tear breakup time, tear film meniscus area, and meibomian gland area were increased. These results suggest that topical diquafosol therapy is effective for patients with obstructive MGD. However, so far, no studies have reported the effect of DQS combined with eyelid hot compress and eyelid gland massage for MGD.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with FBUT<10s；
2. Presence of ocular symptoms with OSDI score≥13；
3. 0<The score of meibum quality or expressibility ≤2；
4. 1/3≤The meibomian drop-out ≤2/3 (meiboscore ≤2)

Exclusion Criteria:

1. patients diagnosed of dry eye with Sjogren syndrome or diabetic mellitus.
2. Patients who wear contact lens during study or accepted refractive surgery within 6 months before screening.
3. Patients who have allergy history or adverse reactions to the experimental drugs or its components.
4. Patients with active ocular inflammation such as infectious keratitis or blepharitis.
5. Patients who had received ocular or system steroids or immunosuppressant 2 weeks before screening.
6. Patients who had received any other experimental drug 2 weeks before screening.
7. Patients with concomitant disease who were considered unable to evaluate efficacy or unlikely to complete the expected course of treatment and follow-up.
8. Pregnant and lactating women, or those planning a pregnancy over the course of the study.
9. Patients judged by the investigator to be unsuitable for the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2022-08-05 (Actual); Primary Completion 2024-05-20 (Estimated); Study Completion 2025-05-20 (Estimated)

PRIMARY OUTCOMES:
The tear fluorescein break-up time changes at 12 weeks from baseline in both groups. | 12 weeks
  The standard TBUT measurement was performed. After 1%fluorescein dye was instilled into the conjunctival sac, the interval between the last complete blink and the appearance of the first corneal black spot in the stained tear film was measured three times and the mean value of the measurements was calculated.

SECONDARY OUTCOMES:
The tear fluorescein break-up time changes at 2 and 4 weeks from baseline in both groups. | 2,4 weeks
  The standard TBUT measurement was performed. After 1%fluorescein dye was instilled into the conjunctival sac, the interval between the last complete blink and the appearance of the first corneal black spot in the stained tear film was measured three times and the mean value of the measurements was calculated.
The CFS changes at 2 ，4 and 12 weeks from baseline in both groups. | 2,4 and 12 weeks
The OSDI changes at 2 ，4 and 12 weeks from baseline in both groups. | 2,4 and 12 weeks
  The dry eye diagnosis flowchart begins with history-taking, risk factors are questioned in suspicious cases, and a screening test such as the Ocular Surface Disease Index (OSDI) Questionnaire is applied.
The lid margin hyperaemia changes at 2 ，4 and 12 weeks from baseline in both groups | 2,4 and 12 weeks
  lid margin hyperaemia：score=0: no or slightly congested conjunctiva at the eyelid margin, no telangiectasis at the opening of the meibomian gland; score=1: conjunctival congestion at the edge of the eyelid, no telangiectasis at the opening of the meibomian gland; score=2: conjunctival congestion at the edge of the eyelid, telangiectasis at the opening of the meibomian gland, and the scope <1/2 eyelid margin; score=3: conjunctival hyperemia at the eyelid margin, telangiectasis at the opening of the meibomian gland, and the range is 1/2 of the eyelid margin.
The LLT changes at 2 ，4 and 12 weeks from baseline in both groups. | 2,4 and 12 weeks
  LLT:LipiView eye surface interferometer The optical interferometry images of the tear film lipid layer are obtained, and the LLT values are automatically obtained according to the color of the images, and the expression of the optical interferometric color units (ICU). 1 ICU stand for 1 nm LLT. LLT is less than or equal to 60nm, and MGD is 90% probable. The device also can record the number of blinks and the proportion of incomplete blinks.
The TMH changes at 2 ，4 and 12 weeks from baseline in both groups. | 2,4 and 12 weeks
  TMH:measured by tear film pattern of Keratograph 5M (Oculus, Wetzlar, Germany) before other invasive procedures. In the tear meniscus measure section of TF pattern, manually measure the tear meniscus height along the middle of lower eyelid with the ruler option after image.
The meiboscore (meibomian gland drop out score) changes at 2 ，4 and 12 weeks from baseline in both groups. | 2,4 and 12 weeks
  The meibomian glands drop out score(Meiboscore): meiboscore=0: without meibomian gland loss on visual inspection of images. meiboscore=1: with meibomian gland area loss of less than one-third of the total area. meiboscore=2: with meibomian gland area loss between one-third and two-thirds of the total area. meiboscore=3: with meibomian gland area loss of more than two-thirds of the total area. Evaluate the upper eyelid and record the score.
The changes of multi-measurement of Meibomian glands by meibography at 4 and 12 weeks from baseline in both groups | 4 and 12 weeks
The changes of corneal sensitivity at 2, 4 and 12 weeks from baseline in both groups. | 2,4 and 12 weeks
  Cornea sensitivity：Cochet-Bonnet: The gold standard for assessing corneal perception. During the perceptual examination, the patient was asked to look forward and the perceptual apparatus acted vertically on the corneal plane. In general, the higher the number recorded, the more sensitive the cornea. Its measurement should be made before other measurements, especially before topical anesthesia is applied, and the results are more reliable. use Cochet-Bonnet to detect the sensitivity of 5 areas of cornea, the up and down of nasal side, central cornea, the up and down of temporal side.
The correlation between the change trend of meiboscore (meibomian gland drop our score)、meibomian glands opening score、meibum expressibility score、meibum quality score、LLT、corneal sensitivity and FBUT、CFS、OSDI. | 12 weeks
meibomian glands opening score changes at 2 ，4 and 12 weeks from baseline in both groups. | 2,4 and 12 weeks
meibum quality score changes at 2 ，4 and 12 weeks from baseline in both groups. | 2,4 and 12 weeks
meibum expressibility score changes at 2 ，4 and 12 weeks from baseline in both groups. | 2,4 and 12 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Zhongshan Ophthalmic Center, Sun Yat-Sen University, Guangzhou, Guangdong, China